CLINICAL TRIAL: NCT02348996
Title: Randomized Study Comparing Analysis With Bioeletric Impedance and Clinical Evaluation to Determine Dry Weight in Hemodialyis Patients
Brief Title: Study Comparing Dryweight Determination in Hemodialysis Patients With Two Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ana Elizabeth Prado Lima Figueiredo (Other)
Responsible Party: Sponsor-Investigator, Ana Elizabeth Prado Lima Figueiredo, Professor, Pontificia Universidade Católica do Rio Grande do Sul
Organization: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AEFDRYWEIGHT
Record Dates: First submitted 2014-12-10; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical assessment (Other): Patients would have dry weight determined by clinical evaluation (blood pressure levels, peripheral edema, pulmonary auscultation and symptoms).
  Interventions: Other: Clinical evaluation
- Bioimpedance (Experimental): Patients would have dry weight determined according to volume status with a body composition monitor (BCM)
  Interventions: Other: Bioimpedance

INTERVENTIONS:
Other: Bioimpedance — status of overhydration determine by BCM once a week to determine dry weight
  Arms: Bioimpedance
Other: Clinical evaluation — Doctors or nurses will evaluate patients on a daily basis and determine dry weight
  Arms: Clinical assessment

SUMMARY:
Adequate control of extracellular volume is a major goal of renal replacement therapy in patients with chronic renal disease. Fluid overload is present in the early stages of chronic kidney disease and contributes significantly to hypertension, arteriosclerosis and high prevalence of left ventricular hypertrophy. These are associated with high rates of morbidity and mortality in this group of patients, rates on dialysis in Brazil is around17.9 % per year. Dry weight during hemodialysis remains a delicate gap between hypervolemia and hypovolemic. Many studies have shown that tight control of post - dialysis weight is related to better outcomes in short term and higher long-term survival. Many methods have been proposed for estimating the hydration status of hemodialysis patients in an objective manner, including ultrasonography of the inferior vena cava and echocardiography. However, these methods are very time-consuming and cumbersome to use in daily practice. In most dialysis centers, the dry weight is evaluated on subjective clinical criteria, with trial and error and time consuming. It was recently introduced in Brazil to monitor body composition by multifrequency bioimpedance, called Body Composition Monitor ( BCM ) manufactured by Fresenius Medical Care. The BCM is a piece of bioimpedance spectrometry using a three compartment model, able to quantify objectively and accurately the extracellular volume and hydration status of each patient by measuring body resistance to an electric current. The procedure is safe, simple and relatively inexpensive. The BCM uses multi-frequency currents (ranging from 5 to 1000 KHz ). The availability of this device evaluation of body composition which assesses the dry weight more efficiently and objectively determine a target to be achieved to prevent left ventricular hypertrophy, hypertension better manage and improve cardiovascular outcomes, motivates us to perform this study. So the goal is to compare the efficacy between bioelectrical impedance analysis and clinical evaluation for suitability of dry weight in hemodialysis patients. A prospective, randomized, crossover study, which will include all chronic renal failure patients on hemodialysis at St. Luke 's Hospital (PUC - RS), including patients with at least three months on HD and over 18 years of age. The expected primary outcome is to achieve greater accuracy in determining the state of hydration and dry weight of these patients.

DETAILED DESCRIPTION:
All patients in the study will undergo a period of prior randomization of a week, where data will be registered such as pre and post blood pressure, average weight gain (delta weight) between sessions and transdialysis complications.

In the first phase, BIA and clinical evaluation to assess blood volume pre-hemodialysis session state in a single assessment will evaluate all patients in the study. The clinical assessment method of dry weight determination includes: patient history in search of signs and symptoms of volume overload, analysis of pre treatment blood pressure, adventitious sounds in pulmonary auscultation among others.

Patients will be randomized in a systematic manner into two groups:

Group A - Clinic Assessment (AC): patients will have dry weight determine by clinical examination, as unit routine, for four weeks. Clinical criteria for dry weight adjustments are: edema, dyspnea, reported shortness of breath, post dialysis blood pressure greater than or equal 140/90 mmHg.

Group B - bioimpedance (BIA): BIA was used to estimate dry weight for four weeks, pre first HD session of the week.

At the end of the first four weeks both groups will be assessed for hydration state, data registered in specific instrument to assess weight gain between sessions, frequency of complications and time to reach dry weight.

After two weeks' interval, wash out, groups would change the method used to assess their dry weight. ( A - BIA and B -CA) After the second phase, all patients had a further evaluation with BIA to assess for hydration state, weight gain between sessions, frequency of complications and time to reach dry weight, all data registered in a specific instrument. Dry weight was achieved by adjustments made in all HD sessions, based on clinical evaluation or BIA. The maximum decrement to achieved dry weight was 500 grams of weight per dialysis session. Nurses did clinical evaluation in both groups.

The unit heath team, nurses and doctors, trained in the methodology used in the research helped determine dry weight.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis patient over 18 years old that accepted to participate

Exclusion Criteria:

* Patients with metal orthopedic implants, cardiac pacemakers, patients with amputated limbs, due to the failure of evaluation of these patients by bioelectrical impedance analysis (BIA) and patients who do not accept participate in the study or decide to leave during the period of study research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in dry weight(DW) status at 10 weeks | DW assessment every dialysis session for 10 weeks
  Volume status would match dry weight and euvolemia

SECONDARY OUTCOMES:
Decreasing adverse events transdialysis | every dialysis session for 10 weeks
  count of number of adverse events during a dialysis session